CLINICAL TRIAL: NCT07045103
Title: A Multicenter Study in Bronchoscopy Combining Stimulated Raman Histology With Artificial Intelligence for Rapid Lung Cancer Detection
Brief Title: A Multicenter Study in Bronchoscopy Combining Stimulated Raman Histology With Artificial Intelligence for Rapid Lung Cancer Detection - The ON-SITE Study
Acronym: ON-SITE
Status: Recruiting | Type: Observational
Sponsor: Invenio Imaging Inc. (Industry)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); University of North Carolina, Chapel Hill (Other); M.D. Anderson Cancer Center (Other); Mayo Clinic (Other); University of California, San Diego (Other); Montefiore Medical Center-Moses-Weiler (Unknown); Corewell Health (Unknown)
Responsible Party: Sponsor
Other Study IDs: INV-01-2022; 1R44CA281581-01 (NIH)
Record Dates: First submitted 2025-06-20; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Lung Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- ON-SITE Patients: Participants must fulfill all of the following criteria in order to be eligible for the study:
  1. The patient or legal guardian is willing and able to understand, sign and date the Ethics committee-approved study specific Informed Consent Form.
  2. The patient is 22 years of age or older.
  3. The patient is scheduled for routinely indicated staging of the mediastinum (EBUS-TBNA) and planned peripheral lung biopsy procedure (peripheral-TBBx/TBNA) with an intermediate to high pretest probability of lung cancer based on clinician suspicion.
  4. The patient can tolerate the clinical procedure as indicated.

SUMMARY:
The ON-SITE study represents a prospective, observational study focused on the training/tuning and pivotal validation of deep learning algorithms that detect cell/tissue morphology suspicious for cancer in biopsies of peripheral lung nodules/masses and mediastinal/hilar lymph nodes imaged with the NIO Laser Imaging System in the procedure room without requiring traditional sample processing.

The study includes four arms based on biopsy location and biopsy modality/tool:

1. Transbronchial forceps biopsy of peripheral lung nodules/masses (peripheral-TBBx)
2. Transbronchial needle aspiration biopsy of peripheral lung nodules/masses (peripheral TBNA)
3. Transbronchial needle aspiration biopsy of mediastinal/hilar lymph nodes (EBUS-TBNA)
4. Transbronchial cryo biopsy of peripheral lung nodules/masses (peripheral-CBx)

ELIGIBILITY:
Inclusion Criteria:

1. The patient or legal guardian is willing and able to understand, sign and date the Ethics committee approved study specific Informed Consent Form.
2. The patient is 22 years of age or older.
3. The patient is scheduled for routinely indicated staging of the mediastinum (EBUS-TBNA) and planned peripheral lung biopsy procedure (peripheral TBBx/TBNA) with an intermediate to high pretest probability of lung cancer based on clinician suspicion.
4. The patient can tolerate the clinical procedure as indicated.

Exclusion Criteria:

1. Patient is a prisoner.
2. The participant, in the judgment of the Investigator, may be inappropriate for the intended study procedures

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for routinely indicated staging of the mediastinum (EBUS-TBNA) and planned peripheral lung biopsy procedure (peripheral TBBx/TBNA) with an intermediate to high pretest probability of lung cancer based on clinician suspicion.
  Patients who meet criteria will be enrolled consecutively from 5 different Hospitals including MD Anderson Cancer Center, University of North Carolina Medical Center, Corewell Health, Montefiore Medical Center, Memorial Sloan Kettering Cancer Center, University of San Diego, Mayo Clinic
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Peripheral TBBx and CBx Co-primary Endpoints | From enrollment to the End of the Procedure.
  Detection of lung cancer in peripheral TBBx and CBx biopsies by NIO image analysis module with non-inferior performance compared to rapid on-site evaluation touch imprint cytology (ROSE-TIC)
Peripheral Lung Transbronchial Fine Needle Aspiration Endpoint | From enrollment to the End of the Procedure.
  Detection of lung cancer in peripheral lung transbronchial needle aspiration by NIO image analysis module with non-inferior performance compared to rapid on-site evaluation (ROSE).
Lymph Node Endobronchial Ultrasound Transbronchial Fine Needle Aspiration Endpoint | From enrollment to the End of the Procedure.
  Determine area-under-the-curve (AUC) of the receiver-operating-characteristic (ROC) of NIO image analysis module for detection of cancer at a lymph-node location.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - UC San Diego, San Diego, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Corewell Health, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - UNC Medical Center, Chapel Hill, North Carolina
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided